CLINICAL TRIAL: NCT00951834
Title: Sunphenon EGCg (Epigallocatechin-Gallate) in the Early Stage of Alzheimer´s Disease
Acronym: SUN-AK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Friedemann Paul, PI, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUN-AK
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer´s Disease; Epigallocatechin-Gallate; Neuroprotection; ADAS-COG; early stage of Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epigallocatechin-Gallate (Experimental): * Months 1-3: 200 mg EGCG/die (200-0-0 mg)
  * Months 4-6: 400 mg EGCG/die (200-0-200 mg)
  * Months 7-9: 600 mg EGCG/die (400-0-200 mg)
  * Months 10-18: 800 mg EGCG/die (400-0-400 mg)
  add-on to Donepezil.
  Interventions: Drug: Epigallocatechin-Gallate
- Placebo (Placebo Comparator): add-on to Donepezil.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epigallocatechin-Gallate — Epigallocatechin-Gallate (EGCG) - Sunphenon EGCg:
  * Months 1-3: 200 mg EGCG/die (200-0-0 mg)
  * Months 4-6: 400 mg EGCG/die (200-0-200 mg)
  * Months 7-9: 600 mg EGCG/die (400-0-200 mg)
  * Months 10-18: 800 mg EGCG/die (400-0-400 mg)
  Other Names: Sunphenon EGCG
  Arms: Epigallocatechin-Gallate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
EGCG has shown a neuroprotective effect in cell-experimental and animal studies. The neuroprotective mechanism of EGCG probably bases - besides the known antioxidant effect - amongst others on the modulation of several signal transduction pathways, the influence on the expression of genes which regulate cell survival resp. programmed cell death, as well as the modulation of the mitochondrial function. In different Alzheimer models EGCG seems to cause an induction of alpha-secretase and the endothelin-converting-enzyme, as well as to prevent the aggregation of beta-amyloid to toxic oligomers through the direct binding to the unfolded peptide.

The investigators therefore expect EGCG to have a positive influence on the course of the Alzheimer´s Disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive dementia characterised by an ongoing loss of memory function and of at least one additional cognitive domain resulting in impairment of daily life functioning. Treatment of diseases such as diabetes mellitus, fractures and cardiovascular diseases is more expensive and complicated in patients with dementia compared to those without. The yearly costs for treatment and care of AD patients in the US are estimated to exceed 100 billion USD. Life expectancy is reported to be about 10 years after establishment of the diagnosis and is significantly reduced compared to non-demented subjects of similar age and socio-economic status.

Age is the most relevant risk factor for AD, followed by genetic factors. Prevalence is less than 1% amongst individuals aged 50-60, but is reported to double every 5 years beyond the age of 60. The prevalence exceeds 30% in the age of 85-90.

The only standard therapy for AD are acetylcholine-esterase inhibitors (AchEI; donepezil, galantamine, rivastigmine). AchEI exhibit a temporary stabilizing mild effect on the progression of AD. Conversion rates from "mild cognitive impairment" to AD do not seem to be beneficially influenced by AchEI. A high percentage of premature study withdrawals owing to adverse events has been observed in AchEI studies published to date. The questionable benefit may further be outweighed by high costs of the AchEI.

Therefore, there is a necessity for the development of more efficacious and less expensive disease-modifying drugs with a better safety and tolerability profile. EGCG is a promising compound which has proven efficacious in AD animal models and which has shown an excellent tolerability in our 18-month clinical trial on Multiple Sclerosis currently being performed at our institution (SuniMS study, NCT00525668).

ELIGIBILITY:
Inclusion Criteria:

* early stage of AD (Diagnosis DSM-IV and NINCDS/ADRDA, Dubois-criteria 2007)
* age 60-100
* MMSE 20-26
* patient lives at home with at least one relative who perform external ratings/assessment
* co-medication with Donepezil (Aricept®, Pfizer Pharma GmbH) with at least 3 months to maximum 6 months of existing stable medication
* maximum of 2 cups of black tea/die, no green tea, not more than > 500 ml/die of grapefruit juice

Exclusion Criteria:

* co-medication with NSAIDs (longterm medication) (ASS is not an exclusion criteria), Gingko- or other natural extracts, other anti-dementiva except of Donepezil
* familial autosomal-dominant inherited AD
* instable medical condition
* other primary psychiatric/neurologic disorders
* missing informed consent
* no readiness to save and refer pseudonym personal data
* hospitalisation due to juridical or legal regulation
* any condition disturbing or making MRI and other measures impossible
* clinically relevant GI-disorders at screening and 1 year before
* clinically relevant lung, infectious, heart or other CNS disorders, clinical or paraclinical suspicion of TBC, history of vascular CNS-disorders at screening and 1 year before
* clinically relevant liver disorders at screening and 1 year before
* clinically relevant functional disorders of liver, kidney or bone marrow defined by following lab values at screening:

  * Marrow dysfunction:

    * HB < 8,5 g/dl
    * WBC < 2,5/nl
    * Thrombocytes < 125/nl
  * Kidney dysfunction:

    * Creatinin-Clearance according to Cockcroft-Gault-Formula: Cl < 110ml/min (male) resp. Cl < 95ml/min (female), from the age of 30 decline of 10ml/min per decade
  * Liver dysfunction:

    * ASAT/ALAT > 3.5 x higher than the upper reference value
    * Bilirubin > 2.0 mg/dl
* known allergy of elements of Sunphenon EGCg or additives of Sunphenon EGCg resp. placebo
* long-term hepatotoxic medication
* current intake of cytochrom P450 3A4-inhibitors or -inductors, such as antimycotics of the azol-type or macrolide-antibiotics
* clinical-anamnestic or paraclinical manifestations suggesting an alcohol or drug abuse
* participation in any clinical trial < 3 months prior to screening or ongoing
* any medical, psychiatric or other condition which might constrain the ability of the patient to understand the informed consent, to give consent, to adhere to the protocol or to accomplish the study
* massive and extended sun exposure

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
ADAS-COG (Score 0-70) (Baseline to treatment) | 18 months

SECONDARY OUTCOMES:
Safety and tolerability of the verum | 18 months
MMSE (Score 0-30) after 18 months compared to baseline | 18 months
Time to hospitalisation and Time to death related to AD | 18 months
Brain atrophy assessed by brain MRI | 18 months
Baseline-ADAS-COG and Baseline-MMSE as covariates | 18 months
CIBIC+ and WHO-QOL-Bref | 18 months
Trail Making Test and MVGT | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, MD, Principal Investigator — Charite University Medicine Berlin, NeuroCure
Locations (3):
- Germany (3):
  - Charite University Medicine Berlin, Berlin
  - Charité Universitätsmedizin Berlin Klinik für Psychiatrie und Psychotherapie, Berlin
  - Klinik für Neurologie, Ulm

REFERENCES:
- See also: Related Info — http://www.neurocure.de